CLINICAL TRIAL: NCT02701660
Title: Remote-controlled Dispensing of Medication and Electronic Monitoring of Adherence in Ambulatory Patients With Opioid Dependency Syndrome and Polypharmacy - a Feasibility Trial
Brief Title: Adherence to Polypharmacy in Patients With Opioid Substitution Therapy Using Electronics
Acronym: APPOSTEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APPOSTEL-1
Record Dates: First submitted 2014-11-25; First posted 2016-03-08 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Substance-Related Disorders
Keywords: Pharmaceutical Care; Adherence; Polypharmacy; e-Health; opioid substitution therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electronic medication dispenser (Experimental): An Automatic Tablet Dispensing and Packaging System is used to repack all solid oral prescription medications for each participant into unit-of-dose pouches. Every participant receives a roll with pouches for 14-28 days loaded into a dispenser installed at their homes. The electronic medication dispenser is a remote controlled, electronic medication management aid reminding the patients with acoustic alerts to take their medication.
  Interventions: Device: electronic medication dispenser (medido)

INTERVENTIONS:
Device: electronic medication dispenser (medido) — Automated dispense of medication through an electronic dispenser
  Other Names: medido

SUMMARY:
Electronic dispensers for polypharmacy are used in home care to assist patients with their medication management and to improve adherence. Opioid dependent patients with substitution therapy often exhibit multiple risk factors for non-adherence. The increase of both the age and associated comorbidities in this population demand for innovative solutions to optimize medication management. The investigators developed a novel medication supply model with an automated electronic medication dispenser to simultaneously assist opioid dependent patients with their medication and objectively monitor their adherence. This study aims to demonstrate the feasibility of the new supply model.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent given
* reading and writing skills in German
* Stable housing situation in the canton of Basel-City and adjacent communities
* Accessibility by phone
* Minimum duration in opioid substitution treatment for 2 months
* Polypharmacy (> 3 solid oral medications)
* Routine monitoring of clinical parameters less than 1 week before inclusion or agreed within 1 week from inclusion
* Insured with Swiss health insurance

Exclusion Criteria:

* opioid substitution treatment with Diacetylmorphine
* > 2 drugs, which can not be packaged in pouches (eg liquids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Taking Adherence (Number of days with correctly dispensed pouches (%) | continuous, up to 24 weeks
  Number of days with correctly dispensed pouches (%)

SECONDARY OUTCOMES:
Timing adherence (number of correctly dispensed pouches within predefined time-frame (%) | continuous, up to 24 weeks
  number of correctly dispensed pouches within predefined time-frame (%)
Patients' specific routine parameters according to condition(s) of participant (composite outcome) | up to 24 weeks
  Individual clinical outcomes, eg blood pressure, blood sugar, HIV count...
Psychological distress | inclusion, week 12, 24, 36
  SCL-90R self-report questionnaire
Quality of Life | inclusion, weeks 3, 6, 9, 12, 15, 18, 21, 24, 36
  SF-12 self-report questionnaire
Satisfaction | week 12, 24, 36
  self-report questionnaire, interview
Instrumental Activities of Daily Living | inclusion, week 12, 24, 36
  Instrumental Activities of Daily Living Scale (Lawton-Brody)
Cognitive Impairment | inclusion, week 12, 24, 36
  Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Hersberger, Prof. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- Outpatient addiction service, University Psychiatric Clinics, Basel, Switzerland